CLINICAL TRIAL: NCT05272748
Title: The Effects of Conventional Exercise Combined With Core Stabilization Exercise by Telerehabilitation on Pain, Postural Control, Functional Level and Fear of Fall in Patients With Hip and/or Knee Osteoarthritis
Brief Title: The Effects of Conventional Exercise Combined With Core Stabilization Exercise by Telerehabilitation in Patients With Hip and/or Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21-90
Record Dates: First submitted 2022-02-28; First posted 2022-03-09 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-03

CONDITIONS: Hip Osteoarthritis; Knee Osteoarthritis
Keywords: hip osteoarthritis; knee osteoarthritis; telerehabilitation; core stabilization
MeSH Terms: conditions — Osteoarthritis, Hip; Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Exercise + Core Stabilization Exercise (Experimental): Conventional exercises and core stabilization exercises will be performed with the telerehabilitation method for 8 weeks. Patients will be contacted via laptop, ipad and phones with cameras, microphones and internet connection. Exercise by telerehabilitation will be implemented with a live connection for the first 4 weeks. In the second 4 week periods, exercise videos will be given to the patients and it will be checked by phone. In addition to the exercises in the conventional exercise group, patients will perform pelvic tilt, lateral bridge, single leg bridge, plank, extremity exercises in the crawling position, abdominal crunch, oblique crunch, dead bug, superman exercise. Exercises will be applied 3 times a week.
  Interventions: Other: Conventional Exercise + Core Stabilization Exercise
- Conventional Exercise (Experimental): Conventional exercises used in the treatment of knee and hip osteoarthritis will be performed by the telerehabilitation method for 8 weeks. Patients will be contacted via laptop, ipad and phones with cameras, microphones and internet connection. Exercise by telerehabilitation will be implemented with a live connection for the first 4 weeks. In the second 4 week periods, exercise videos will be given to the patients and it will be checked by phone. Terminal knee extension, straight leg raise, heel slide, adductor isometric, bridge, mini squat, heel raise, lunge, range of motion and stretching exercises for lower extremities will be performed by the patients. Exercises will be applied 3 times a week.
  Interventions: Other: Conventional Exercise

INTERVENTIONS:
Other: Conventional Exercise + Core Stabilization Exercise — Before and after the treatment, patients' pain, postural control (static and dynamic balance), functional level and fear of falling will be evaluated. In addition to the exercises in the conventional exercise group, patients will perform pelvic tilt, lateral bridge, single leg bridge, plank, extremity exercises in the crawling position, abdominal crunch, oblique crunch, dead bug, superman exercise. Exercises will be applied 3 times a week.
  Arms: Conventional Exercise + Core Stabilization Exercise
Other: Conventional Exercise — Before and after the treatment, patients' pain, postural control (static and dynamic balance), functional level and fear of falling will be evaluated. Terminal knee extension, straight leg raise, heel slide, adductor isometric, bridge, mini squat, heel raise, lunge, range of motion and stretching exercises for lower extremities will be performed by the patients. Exercises will be applied 3 times a week.
  Arms: Conventional Exercise

SUMMARY:
Age-related hip and knee osteoarthritis is the leading cause of pain and locomotor problems worldwide. There is no definitive solution in the treatment of hip and knee osteoarthritis. In the guidelines of the American Rheumatology Association, pharmacological and non-pharmacological treatment methods are recommended for the treatment of hip and knee osteoarthritis. The effectiveness of different exercise programs for the periarticular muscles in hip and knee osteoarthritis has been proven, but there is no consensus on the superiority of exercise protocols over each other. With the increase in home isolation of individuals due to the COVID-19 pandemic, telerehabilitation applications have gained popularity.In the literature, there is a need for studies investigating the effectiveness of core stabilization exercises in patients with hip and knee osteoarthritis. Therefore, our study will help develop alternative exercises for individuals with hip and knee osteoarthritis. In the literature, there is no study investigating the effectiveness of core stabilization exercises applied with the telerehabilitation method in patients with knee osteoarthritis and comparing them with conventional exercise. According to the data to be obtained as a result of the study, the use of core stabilization exercises in the treatment of hip and knee osteoarthritis will contribute to the literature as an alternative exercise method. The application of these exercises with the telerehabilitation method in the treatment of hip and knee osteoarthritis will highlight new studies in the literature as a unique methodology. Thus, it will contribute to the development of cost-effective rehabilitation methods in the treatment of hip and knee osteoarthritis.

The hypotheses of this study are as follows:

H0:There is no difference between the effects of combined exercise with telerehabilitation (conventional exercise + core stabilization exercise) and the effects of conventional exercise in the treatment of hip and/or knee osteoarthritis.

H1:Combined exercise with telerehabilitation application (conventional exercise + core stabilization exercise) is more effective than conventional exercise in the treatment of hip and/or knee osteoarthritis.

Main Purpose: To compare the effects of conventional exercise and core stabilization exercises by telerehabilitation on pain, postural control, functional level, and fear of falling in patients with hip and/or knee osteoarthritis.

Secondary Purposes:

* To evaluate the effects of core stabilization exercises on pain, postural control, functional level, fear of falling in female patients with hip and/or knee osteoarthritis.
* To evaluate the effectiveness of telerehabilitation exercise in female patients with hip and/or knee osteoarthritis.
* To determine the possible limitations that may be encountered in the application of exercise by telerehabilitation in female patients with hip and/or knee osteoarthritis and to provide appropriate conditions for the patients.

ELIGIBILITY:
Inclusion Criteria:

* Woman
* 40 years or older
* Diagnosed with primary hip and/or knee osteoarthritis as a result of radiological and clinical examination
* Informed written consent

Exclusion Criteria:

* Using an assistive device
* Prior orthopedic surgery of the knee and hip
* Intra-articular injection of the knee in the last 3 months
* Clinical or radiological meniscus, cartilage and/or ligament problem
* Severe physical trauma in the past 3 months
* Severe psychological trauma in the past 3 months
* Arterial and venous circulation disorder
* Presence of skin lesions on and around the knee joint
* Presence of neuromuscular disease and/or neurological deficit
* Presence of vertigo, diabetes mellitus, hearing and vision problems
* Not having the technologies to access telerehabilitation services

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only Female Participants
Enrollment: 23 (Actual)
Dates: Start 2022-03-16 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-06-11 (Actual)

PRIMARY OUTCOMES:
Numerical Rating Scale (NRS) | Change from Baseline NRS Score at 8 weeks
  Numerical Rating Scale (NRS) is used for the evaluation of pain intensity. This 11-point scale is used to measure the severity of pain between 0 and 10 points. In the scale, there are numbers between 0 and 10 arranged horizontally, with 0: "No pain", 10: "Unbearable pain".
Berg Balance Scale (BBS) | Change from Baseline BBS Score at 8 weeks
  Berg Balance Scale (BBS) examines both static and dynamic balance functions. BBS consists of 14 items and evaluates the ability of individuals to maintain their balance during activities. Each section is scored between 0 and 4 as 0: "Activity Not Completed", 4: "Activity Independent" completed.
Timed Up and Go Test (TUG) | Change from Baseline TUG Score at 8 weeks
  Timed Up and Go Test (TUG) is used for the evaluation of functional level. After the patient rested for 15 seconds in a back-supported chair, the test is started with the command "start". The patient is asked to get up from the chair without support from the hands and walk the marked 3-meter track, as quickly as possible, but without running, at his own pace, and sit back on the chair, and the elapsed time is recorded in seconds. A trial was made for the patient to learn the test, and then the test was repeated 3 times and the average time was recorded.
Knee Injury and Osteoarthritis Outcome Score - Physical Function Short Form (KOOS-PS) | Change from Baseline KOOS-PS Score at 8 weeks
  Knee Injury and Osteoarthritis Outcome Score - Physical Function Short Form (KOOS-PS) is used for the evaluation of functional level in patients with knee osteoarthritis. Each question is answered using a score of 0-4 (0: "None" - 4: "Extreme") with five answer options.
Hip Disability and Osteoarthritis Outcome Score - Physical Function Short Form (HOOS-PS) | Change from Baseline HOOS-PS Score at 8 weeks
  Hip Disability and Osteoarthritis Outcome Score - Physical Function Short Form (HOOS-PS) is used for the evaluation of functional level in patients with hip osteoarthritis. Each question is answered using a score of 0-4 (0: "None" - 4: "Extreme") with five answer options.
The Falls Efficacy Scale International (FES-I) | Change from Baseline FES-I Score at 8 weeks
  The Falls Efficacy Scale International (FES-I) is used for the evaluation of fear of fall. Each question is answered using a range of 1-4 points (1: "Not at all concerned" - 4: "Very concerned") with four answer options.

CONTACTS AND LOCATIONS:
Overall Officials: Zuhal Didem Takinacı, Asst. Prof., Principal Investigator — Saglik Bilimleri Universitesi; İlknur Aktaş, MD., Prof., Principal Investigator — Sağlık Bilimleri Üniversitesi Fatih Sultan Mehmet Eğitim Ve Araştırma Hastanesi
Locations (2):
- Turkey (Türkiye) (2):
  - Sağlık Bilimleri University, Istanbul
  - Sağlık Bilimleri Üniversitesi Fatih Sultan Mehmet Eğitim Ve Araştırma Hastanesi, Istanbul

IPD SHARING:
Plan to Share IPD: No